CLINICAL TRIAL: NCT02354560
Title: Erythromycin Treatment for Readthrough of APC Gene Stop Codon Mutation in Familial Adenomatous Polyposis-protocol is Identical to Study No. 0519-10-TLV- Minors' Adjusted Version
Brief Title: Erythromycin Treatment for Readthrough of APC Gene Stop Codon Mutation in Familial Adenomatous Polyposis-minors' Adjusted Version
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: michal roll (Other Government)
Responsible Party: Sponsor-Investigator, michal roll, director, R&D Division, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0377-14-TLV
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: FAP-Familial Adenomatous Polyposis
Keywords: Erythromycin; Familial Adenomatous Polyposis (FAP); APC gene; nonsense mutations
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythromycin (Experimental): Oral treatment with Erythromycin 250-500mg (will be determined according to body weight) twice a day.
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin — Oral Treatment with Erythromycin 250-500mg, twice daily, for 16 weeks.Exact dose is subjected to body weight and will be determined by the study's pediatrician.

SUMMARY:
Colorectal cancer (CRC) is a leading cause for cancer related mortality in the western world with a lifetime risk of 6%. Etiology is complex, while genetic background significantly affects the risk. Around one third of all genetic disorders as well as most cases of Familial Adenomatous Polyposis (FAP) and a large proportion of all sporadic CRC cases occur as a result of premature nonsense mutations (creating a stop codon) in an individual's adenomatous polyposis coli (APC) gene. Nonsense mutations are single-point alterations in the DNA that prematurely halt the protein translation process, producing a shortened, nonfunctional protein. In many of these cases, if the cell can be 'persuaded' to ignore the premature stop codon signal, the resulting protein may be able to ameliorate or stop the disease.

Recently, members of the aminoglycoside family of antibiotics have been found to induce ribosomal read-through of nonsense mutations, leading to expression of a full length, functional protein. Investigators have recently shown that members of the aminoglycoside and macrolide antibiotic families can induce read-through of the nonsense mutations in the APC gene and lead to reduced oncogenic phenotypes in CRC cells and in different mice models.

The aim of this project is to determine the ability of the macrolide antibiotic-erythromycin to induce read-through of the nonsense mutations in the APC gene and to induce expression of a full length, functional APC protein in patients suffering from FAP and to tests its effect on adenoma number and size and on desmoid tumors in these patients. The future goal is to maximize the effect of stop-codon suppressors on APC while minimizing side effects.

In this study investigators will select FAP patients which carry APC nonsense mutations, treat them with erythromycin PO for 4-6 months and examine colonic and duodenal adenomas as well as abdominal desmoid tumors, that will be documented before during and after treatment. In parallel, investigators will test polyp, adenoma and desmoid tissue samples as well as blood samples from these patients for changes in expression levels of the APC protein and related oncogenic markers.

Suppression of nonsense mutations within the APC gene should be of benefit for patients suffering from FAP, attenuated FAP or multiple adenomas and for patients with advanced or diffuse CRC. Furthermore, given the rapid progress being made in the identification of different nonsense mutations in human genes that lead to mostly un-curable disease, the identification of clinically approved compounds that suppress nonsense mutations and that can be administered long-term without significant side effects would open new venues in the treatment of genetic human diseases that arise from pre-mature stop codons in important coding sequences.

Immediate goal: establish the ability of erythromycin to read-through APC nonsense mutation in FAP patients. The read-through effect of erythromycin will be clinically tested by counting and measuring the number and size of both colonic and duodenal adenomas before and over treatment and by measuring the size of known desmoid tumors. Samples of the adenomas and desmoid tumors will be tested by western blot, immunofluorescence and immunohistochemistry for restoration of APC expression and changes in oncogenic markers. These experiments should be conducted within 6 month.

Long term objective:

1. Determine the lowest dose of erythromycin that can inhibit growth of colonic neoplasia and CRC in patients expressing a truncated APC protein due to nonsense mutations.
2. Examine the ability of a panel of additional macrolide antibiotics to induce APC nonsense mutation suppression using in-vitro methods. Investigators will focus on macrolide antibiotics that are currently in clinical use and are administrated for long terms. These objectives should take around 6 month and will be conducted in parallel.

ELIGIBILITY:
Inclusion Criteria:

* ages: 10-17 years old.
* A lack of known sensitivity to ERYTHROMYCIN or other macrolide.
* at the relevant subgroup - existence of polyps in the colon or Ileo-anal pouch that classified as adenomas and the size isn't bigger than 10 mm and there's no high grade dysplasia and that not yet need immediate resection of the colon rectal but just a surveillance.
* In the relevant subgroup- existence of polyps in the duodenum that do not require surgery and aren't bigger than 10 mm and with out high grade dysplasia.
* In the relevant subgroup- a tumor that classified as stomach or pelvic desmoid that not yet need immediate resection and which can be measured by ultrasound or MRI.

Exclusion Criteria:

* below 10 years old or above 18 years old.
* sensitivity to ERYTHROMYCIN or other macrolide.
* Ileo-anal pouch without adenomas.
* existence of polyps that are classified as adenomas which are bigger than 10 mm and/or with histological of high grade dysplasia.
* Taking medicines that have interactions with ERYTHROMYCIN such as: Carbamazepine, Cyclosporine, barbiturate, PHENYTOIN, Disopyramide, Lovastatin, Bromocriptine: it is recommended to keep careful attention over their Concentrations in the blood and to match the dose.
* significant personal of familial history of ventricular arrhythmia and/or Long QT interval per ECG, or consumption of drugs that may cause prolonged QT.
* Recruitment of children whom suffer from FAP in addition to other diseases is subject to a joint decision of the PI and the study pediatrician.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in number of adenomas measured by upper endoscopy | After 8,16 weeks and 12 months
  Change in number of adenomas from baseline will be measured by endoscopic and histological evaluation. response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment.
Evaluation of changes in size of adenomas measured by lower endoscopy | After 8,16 weeks and 12 months
  Change in number of adenomas from baseline will be measured by endoscopic and histological evaluation. response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment.
Evaluation of changes in size of desmoid tumors | At the begining of the trial (before treatment) and at the end of the treatment (after 4-6 months)
  Desmoids imaging (US or CT or MRI) will be performed to determine the size at the begining of the study and to evaluate the change from baseline after 4-6 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Revital Kariv, MD, Study Director — Department of Gastroenterol Tel Aviv Medical Center, Sackler Faculty of Medicine, Tel Aviv University.; Rina Rosin-Arbeseld, Ph.D, Study Director — Department of Anatomy Sackler Faculty of Medicine, Tel Aviv University.

REFERENCES:
- [Background] Smith KJ, Johnson KA, Bryan TM, Hill DE, Markowitz S, Willson JK, Paraskeva C, Petersen GM, Hamilton SR, Vogelstein B, et al. The APC gene product in normal and tumor cells. Proc Natl Acad Sci U S A. 1993 Apr 1;90(7):2846-50. doi: 10.1073/pnas.90.7.2846. PMID 8385345
- [Background] Miyoshi Y, Nagase H, Ando H, Horii A, Ichii S, Nakatsuru S, Aoki T, Miki Y, Mori T, Nakamura Y. Somatic mutations of the APC gene in colorectal tumors: mutation cluster region in the APC gene. Hum Mol Genet. 1992 Jul;1(4):229-33. doi: 10.1093/hmg/1.4.229. PMID 1338904
- [Background] Jasperson KW, Tuohy TM, Neklason DW, Burt RW. Hereditary and familial colon cancer. Gastroenterology. 2010 Jun;138(6):2044-58. doi: 10.1053/j.gastro.2010.01.054. PMID 20420945
- [Background] Nieuwenhuis MH, Mathus-Vliegen EM, Baeten CG, Nagengast FM, van der Bijl J, van Dalsen AD, Kleibeuker JH, Dekker E, Langers AM, Vecht J, Peters FT, van Dam R, van Gemert WG, Stuifbergen WN, Schouten WR, Gelderblom H, Vasen HF. Evaluation of management of desmoid tumours associated with familial adenomatous polyposis in Dutch patients. Br J Cancer. 2011 Jan 4;104(1):37-42. doi: 10.1038/sj.bjc.6605997. Epub 2010 Nov 9. PMID 21063417
- [Background] Zilberberg A, Lahav L, Rosin-Arbesfeld R. Restoration of APC gene function in colorectal cancer cells by aminoglycoside- and macrolide-induced read-through of premature termination codons. Gut. 2010 Apr;59(4):496-507. doi: 10.1136/gut.2008.169805. Epub 2009 Dec 1. PMID 19951906
- [Background] Lai CH, Chun HH, Nahas SA, Mitui M, Gamo KM, Du L, Gatti RA. Correction of ATM gene function by aminoglycoside-induced read-through of premature termination codons. Proc Natl Acad Sci U S A. 2004 Nov 2;101(44):15676-81. doi: 10.1073/pnas.0405155101. Epub 2004 Oct 21. PMID 15498871
- [Background] Wilschanski M, Yahav Y, Yaacov Y, Blau H, Bentur L, Rivlin J, Aviram M, Bdolah-Abram T, Bebok Z, Shushi L, Kerem B, Kerem E. Gentamicin-induced correction of CFTR function in patients with cystic fibrosis and CFTR stop mutations. N Engl J Med. 2003 Oct 9;349(15):1433-41. doi: 10.1056/NEJMoa022170. PMID 14534336
- [Background] Kerem E, Hirawat S, Armoni S, Yaakov Y, Shoseyov D, Cohen M, Nissim-Rafinia M, Blau H, Rivlin J, Aviram M, Elfring GL, Northcutt VJ, Miller LL, Kerem B, Wilschanski M. Effectiveness of PTC124 treatment of cystic fibrosis caused by nonsense mutations: a prospective phase II trial. Lancet. 2008 Aug 30;372(9640):719-27. doi: 10.1016/S0140-6736(08)61168-X. Epub 2008 Aug 20. PMID 18722008
- [Background] West NJ, Clark SK, Phillips RK, Hutchinson JM, Leicester RJ, Belluzzi A, Hull MA. Eicosapentaenoic acid reduces rectal polyp number and size in familial adenomatous polyposis. Gut. 2010 Jul;59(7):918-25. doi: 10.1136/gut.2009.200642. Epub 2010 Mar 26. PMID 20348368
- [Background] Lips DJ, Barker N, Clevers H, Hennipman A. The role of APC and beta-catenin in the aetiology of aggressive fibromatosis (desmoid tumors). Eur J Surg Oncol. 2009 Jan;35(1):3-10. doi: 10.1016/j.ejso.2008.07.003. Epub 2008 Aug 21. PMID 18722078
- [Result] Markowitz SD, Bertagnolli MM. Molecular origins of cancer: Molecular basis of colorectal cancer. N Engl J Med. 2009 Dec 17;361(25):2449-60. doi: 10.1056/NEJMra0804588. No abstract available. PMID 20018966